CLINICAL TRIAL: NCT04647045
Title: An Evaluation of Cultured Milk Drink on Immune Status of Patients With Constipation Predominant Irritable Bowel Syndrome
Brief Title: An Evaluation of Cultured Milk Drink on Immune Status of Patients With Irritable Bowel Syndrome: Constipation Predominant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Malaysia (Other)
Collaborators: COTRA ENTERPRISES SDN BHD, MALAYSIA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: UKM PPI/111/8/JEP-2017-206
Record Dates: First submitted 2020-11-20; First posted 2020-11-30 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Irritable Bowel Syndrome With Constipation
Keywords: Irritable bowel syndrome; cultured milk drinks; interleukin-6; interleukin-8; tumor necrosis factor-alpha
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: A randomized single-blind case controlled trial was performed in patients who were diagnosed with constipation-predominant irritable bowel syndrome. Each recruited participant was given three bottles of 125 ml cultured milk drink containing 109 cfu Lactobacillus acidophilus LA-5 and Lactobacillus paracasei L. CASEI-01 consumed daily for 30 days. At pre- and post-30-day consumption, fecal pH, ITT, clinical symptoms, IL-6, IL-8 and TNF-α levels were assessed.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IBS-C group (Active Comparator): 77 constipation-predominant IBS were given three bottles of 125 ml cultured milk drink daily for 30 days
  Interventions: Dietary Supplement: Cultured milk drink
- Non-IBS group (Other): 88 non-IBS subjects (healthy individuals) were given similar probiotics for 30 days.
  Interventions: Dietary Supplement: Cultured milk drink

INTERVENTIONS:
Dietary Supplement: Cultured milk drink — Each bottle contains 109 cfu Lactobacillus acidophilus LA-5 and Lactobacillus paracasei L. CASEI-01. In each 100 ml unit, it contains 4.06 g of fructose, 4.14 g of glucose, 0.29 g of sucrose, less than 0.1 g of maltose and 1.35 g of lactose.
  Other Names: Vitagen

SUMMARY:
Our previous work on the use of probiotics improved the clinical symptoms in irritable bowel syndrome with constipation-predominant. This study would like to explore further use of probiotics in the immune system of the patients with irritable bowel syndrome.

DETAILED DESCRIPTION:
This is a case control study involving participants who fulfilled the Rome III criteria for constipation-predominant irritable bowel syndrome. The patients were recruited from the Gastroenterology clinic at Universiti Kebangsaan Malaysia Medical Centre, Kuala Lumpur. A total of 165 participants were recruited based on probability (power) of 0.8 and Type I error was set at 0.05.

The investigators included healthy participants above 18 years old. Those less than 18 years old; constipation due to other medical illnesses such as diabetes mellitus, inflammatory bowel disease, hypothyroidism, colorectal cancer, neurological diseases, major depression, lactose intolerance, pregnancy, breastfeeding women and must not be on chronic opioids or anti- depressants were excluded. Participants must not consume any antibiotics, probiotic, prebiotic, symbiotic and/or laxatives less than two weeks before recruitment.

Participants were required to consume three bottles of 125 ml cultured milk drink daily for 30 days. Each bottle contains 10^9 cfu Lactobacillus acidophilus LA-5 and Lactobacillus paracasei L. CASEI-01. In each 100 ml unit, it contains 4.06 g of fructose, 4.14 g of glucose, 0.29 g of sucrose, less than 0.1 g of maltose and 1.35 g of lactose. Cold chain was maintained below 10°C during storage, transportation and distribution. Prior to consumption of the cultured milk drinks, fecal and blood samples from the participants were obtained to determine their baseline fecal pH and serum cytokines level respectively. Each of the participants answered a food frequency questionnaire to assess their dietary profile (data are not presented in this paper) and the Garrigues Questionnaire to evaluate their clinical symptoms and physical activity. The same parameters were taken following 30 days of cultured milk drinks' consumption.

ELIGIBILITY:
Inclusion Criteria:

* Do not fulfil the Rome III criteria for irritable bowel syndrome

Exclusion Criteria:

* constipation due to other medical illnesses such as diabetes mellitus, inflammatory bowel disease, hypothyroidism, colorectal cancer, neurological diseases, major depression, lactose intolerance, pregnancy, breastfeeding women and must not be on chronic opioids or anti- depressants. Participants must not consume any antibiotics, probiotic, prebiotic, symbiotic and/or laxatives less than two weeks before recruitment.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 165 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Serum cytokine level | 30 days
  Serum cytokine was determined using ELISA method at day 0 and day 30.

SECONDARY OUTCOMES:
Intestinal transit time | 30 days
  Intestinal transit time was determined using red carmine capsule prior to the consumption of probiotics.
Fecal pH | 30 days
  Litmus pH paper was used to determine fecal pH at day 0 and day 30
Constipation related symptoms | 30 days
  Garrigues Questionnaire was used to assess the symptoms at day 0 and day 30. The questions are asked to each participant in the form of 'yes' or 'no'. The symptoms are straining during defecation, passing hard stool, number of bowel movements per week and incomplete emptying sensation after bowel movement. The results were reported as % of patients having the listed symptoms at pre- and post-intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Norfilza M Mokhtar, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No
The investigators are bound to the Institutional Review Board Universiti Kebangsaan Malaysia Medical Research Ethics Committee rules and regulations where recruited patients identity and data are kept confidential and will only be allowed to access by the research team.